CLINICAL TRIAL: NCT00287547
Title: Phase II Randomized, Double-Blind, Placebo-Controlled Study of BMS-188667 (CTLA4Ig) in Patients With Psoriasis Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-005
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-04

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Abatacept

INTERVENTIONS:
Drug: CTLA4Ig / Abatacept

SUMMARY:
The purpose of this study is to assess the safety, pharmacokinetics and clinical activity and immunogenicity of BMS-188667 (CTLA4Ig) in subjects with psoriasis vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis and documentation of a history of stable psoriasis vulgaris of at least 6 months duration.
* vulgaris total body surfae area involvement of at least 10%
* Failure for toxicity and/or inefficacy of at least one standard anti- psoriatic therapy including topical treatment, phototherapy, photochemotherapy, methotrexate, cyclosporin A or etretinate.

Exclusion Criteria:

* Male and female subjects who are not willing to receive adequate counseling and exercise adequate contraceptive measures with enrolle on study.
* Functional class (V (ACR) RA or amyloidosis)
* Active vasculitis (except for subcutaneous rheumatoid nodules).
* Subjects with a history of asthma, angioedema or anaphylaxis.
* Subjects with evidence of active or latent bacterial or viral invedtions.
* Subjects with a history or malignancy (except basal cell or superficial squamous cell skin carcinoma).
* body weight > 100 kg (or 220 lbs.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144
Dates: Start 1997-03; Primary Completion 1998-01 (Actual); Study Completion 1998-01 (Actual)

PRIMARY OUTCOMES:
Using the Psoriasis Disablity Index (PDI) and other assessment tools to determine if the patient's psoriasis improved or worsened over the course of the study.

SECONDARY OUTCOMES:
Safety and immunogenicity; pharmacodynamic and PK; Percent reduction in PASI, PASI component scores and Total Body Surface Area; Clinical response kinetics; clinical relapse kinetics; physician global assessment; psoriasis disability index.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Local Institution, San Diego, California
  - Local Institution, Chicago, Illinois
  - Local Institution, Boston, Massachusetts
  - Local Institution, Ann Arbor, Michigan
  - Local Institution, New Brunswick, New Jersey
  - Local Institution, Portland, Oregon
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Dallas, Texas
  - Local Institution, Salt Lake City, Utah
  - Local Institution, Burlington, Vermont